CLINICAL TRIAL: NCT00806013
Title: Study the Effects of CYP2C9 and CYP2C19 Polymorphisms on the Pharmacokinetics and Pharmacodynamics of Glipizide in Healthy Chinese Subject
Brief Title: Study the Effects of CYP2C Polymorphisms on the Pharmacokinetics and Pharmacodynamics of Glipizide
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Other Study IDs: SIMM-080601
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-12

CONDITIONS: Healthy
Keywords: genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The whole blood samples of each person are stored at -80℃.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: CYP2C9*1/*1 and CYP2C19*1/*1 alleles carrier
- 2: CYP2C19 PMs (CYP2C19*2/*2, CYP2C19*2/*3 or CYP2C19*3/*3)
- 3: CYP2C9*1/*3 and CYP2C19*1/*1 alleles carrier

SUMMARY:
The aims of this study were to investigate the effects of CYP2C9 and CYP2C19 polymorphisms on the pharmacokinetics and pharmacodynamics of glipizide in healthy Chinese subjects.

DETAILED DESCRIPTION:
Compared with CYP2C19, CYP2C9 polymorphism appears to have a dominant role in glipizide pharmacokinetics and pharmacodynamics in vivo. This indicated that dose adjustment based on CYP2C9 genotype may improve antidiabetic treatment.

ELIGIBILITY:
Inclusion Criteria:

* nonsmokers and in good health

Exclusion Criteria:

* family history of diabetes mellitus
* taking any drug, alcohol, foods containing caffeine, or grapefruits and juice before study

Ages: 21 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male Chinese subjects with different geontype of CYP2C9 and CYP2C19 were enrolled in this study. They are divided into three groups by different geontype.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-08; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Tan, Principal Investigator — Shanghai Institute of Materia Medica, Chinese Academy of Sciences
Locations (1):
- The second hospital to Liaoning University of TCM, Shenyang, Liaoning, China

REFERENCES:
- See also: Our organization — http://english.simm.cas.cn/
- See also: Chinese Academy of Sciences — http://english.cas.cn/
- See also: Liaoning University of TCM — http://www.lnutcm.edu.cn/en/